CLINICAL TRIAL: NCT01044225
Title: CeCil: A Randomized, Non-comparative Clinical Trial of the Effect of Radiation Therapy Plus Temozolomide Combined With Cilengitide or Cetuximab on the 1-year Overall Survival of Patients With Newly Diagnosed MGMT-promoter Unmethylated Glioblastoma
Brief Title: Effect of Radiation Therapy Plus Temozolomide Combined With Cilengitide or Cetuximab on the 1-year Overall Survival of Patients With Newly Diagnosed MGMT-promoter Unmethylated Glioblastoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Results of the phase III RTOG0525 trial made the manufacturer of cilengitide decide to end their support to the trial
Sponsor: Bart Neyns (Other)
Responsible Party: Sponsor-Investigator, Bart Neyns, MD PhD, Universitair Ziekenhuis Brussel
Organization: Universitair Ziekenhuis Brussel (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-012324-83
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Glioblastoma
Keywords: newly diagnosed glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Cetuximab; Cilengitide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cilengitide EMD 121974 (Active Comparator): A dose of 2000 mg by iv administration 2 weekly.
  Interventions: Drug: Cilengitide EMD 121974
- Cetuximab (Active Comparator): An initial dose of 400 mg/m² IV over 2 hours and followed by a weekly dose of 250 mg/m² over 1 hour.
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — An initial dose of 400 mg/m² IV over 2 hours and followed by a weekly dose of 250 mg/m² over 1 hour.
  Arms: Cetuximab
Drug: Cilengitide EMD 121974 — A dose of 2000 mg by IV administration 2 weekly.
  Arms: Cilengitide EMD 121974

SUMMARY:
The investigators propose to conduct a multicenter, open-label, randomized, phase II study in patients with newly diagnosed glioblastoma (CeCil). Patients should meet all eligibility criteria for the CENTRIC phase III trial at the exception that no MGMT-promoter methylation could be demonstrated. The treatment backbone in both study arms will consist of postoperative radiation therapy with concomitant daily temozolomide, followed by 6 cycles of temozolomide according to a 21 out of 28 days regimen (as in the experimental arm of the RTOG 0525 / EORTC 26052-22053 phase III study). In study arm (A) Cilengitide (at a dose of 2000 mg by iv administration, 2x/week) will be added to this backbone while in the second study arm (B), Cetuximab will be added (at an initial dose of 400 mg/m² administered by intravenous infusion over 2 hours and followed by a weekly dose of 250 mg/m² iv over 1 hours). In both study arms, treatment will be administered for 52 consecutive treatment weeks. The 1-year overall survival (1y-OS) following randomization will serve as the primary endpoint in both study arms.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Newly diagnosed histologically proven supratentorial glioblastoma (World Health Organization [WHO] Grade IV, including glioblastoma subtypes, e.g. gliosarcoma).
3. Tumor tissue specimens from the glioblastoma surgery or open biopsy (FFPE block) must be available for MGMT gene promoter status analysis and central pathology review and must have been submitted as part of the screen procedure for the CENTRIC phase III study
4. MGMT gene promoter status determined as NOT methylated during the screen procedure for the CENTRIC phase III study
5. Males or females ≥18 years of age.
6. Interval of ≥2 weeks but ≤7 weeks after surgery or biopsy before first administration of study treatment.
7. Available post-operative Gd-MRI performed within 48 hours after surgery
8. Stable or decreasing dose of steroids for 5 days prior to randomization.
9. Eastern Cooperative Oncology Group performance score (ECOG PS) of 0-1.
10. Meets one of the following recursive partitioning analysis (RPA) classifications:

    * Class III (Age <50 years and ECOG PS 0).
    * Class IV (meeting one of the following criteria: a) Age <50 years and ECOG PS 1 or b) Age ≥50 years, underwent prior partial or total tumor resection, Mini Mental State Examination [MMSE] ≥27).
    * Class V (meeting one of the following criteria: a) Age ≥50 years and underwent prior partial or total tumor resection, MMSE <27 or b) Age ≥50 years and underwent prior open tumor biopsy only).
11. Laboratory values

    * Absolute neutrophil count 1500/mm3.
    * Platelets 100,000/mm3.
    * Creatinin 1.5 x upper limit of normal (ULN) or creatinine clearance rate 60 mL/min.
    * Hemoglobin 10 g/dL.
    * Total bilirubin 1.5 x the ULN.
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) 2.5 x ULN (except when attributable to anticonvulsants).
    * Alkaline phosphatase 2.5 x ULN.
    * Prothrombin time (PT) international normalized ratio (INR) and partial thromboplastin time (PTT) within normal limits.

Exclusion Criteria:

1. Prior chemotherapy within the last 5 years.
2. Prior RT of the head.
3. Receiving concurrent investigational agents or has received an investigational agent within the past 30 days prior to the first dose of Cilengitide.
4. Prior systemic anti-angiogenic therapy.
5. Placement of Gliadel® wafer at surgery.
6. Planned surgery for other diseases (e.g. dental extraction).
7. History of recent peptic ulcer disease within 6 months of enrollment.
8. History of malignancy. Subjects with curatively treated cervical carcinoma in situ or basal cell carcinoma of the skin, or subjects who have been free of other malignancies for 5 years are eligible for this study.
9. History of coagulation disorder associated with bleeding or recurrent thrombotic events.
10. Clinically manifest myocardial insufficiency or history of myocardial infarction during the past 6 months; or uncontrolled arterial hypertension.
11. Inability to undergo Gd-MRI.
12. Concurrent illness, including severe dermatological conditions or infection, which may jeopardize the ability of the subject to receive the procedures outlined in this protocol with reasonable safety.
13. Subject is pregnant or is currently breast-feeding, anticipates becoming pregnant/ impregnating their partner during the study or within 6 months after study participation, or subject does not agree to follow acceptable methods of birth control, such as hormonal contraception, intra-uterine pessary, condoms or sterilization, to avoid conception during the study and for at least 6 months after receiving the last dose of study treatment.
14. Current alcohol dependence or drug abuse.
15. Known hypersensitivity to the study treatment.
16. Legal incapacity or limited legal capacity.
17. Presence of any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
18. Signs and symptoms suggestive of transmissible spongiform encephalopathy, or family members who suffer(ed) from such.
19. Treatment with prohibited concomitant medication as defined in Section

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
the 1 year overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bart Neyns, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (6):
- Belgium (6):
  - Onze-Lieve-Vrouwziekenhuis, Aalst, Aalst
  - ZNA Middelheim, Antwerp, Antwerpen
  - GHdC Charleroi, Charleroi, Charleroi
  - ZOL Campus Sint-Jan, Genk
  - UZ Gent, Ghent
  - UCL de Mont-Godinne, Yvoir